CLINICAL TRIAL: NCT05646251
Title: Intra-procedural Transthoracic EChocardiogram to Facilitate LBBAP
Brief Title: Intra-procedural Transthoracic EChocardiogram to Facilitate Left Bundle Branch Area Pacing (LBBAP)
Acronym: EC-LBBAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0917
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: Twenty patients will undergo intraprocedural transthoracic echocardiogram via standard practices. An additional 10 patients will undergo intraprocedural transthoracic echocardiogram using a hand-held ultrasound device. The study team will retrospectively identify 30 consecutive previous patients who satisfy inclusion and exclusion criteria (control patients). The study team will compare the difference in procedural success between Case and Control patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- EC-LBBAP Participant (Experimental): A heart ultrasound will be used during a pacemaker implant procedure
  Interventions: Device: Heart Ultrasound
- Control participant (No Intervention): A pacemaker will be implanted using routine protocol. This is retrospectively collected; patients are not actively enrolled in this arm.
- ECLBBAP handheld participant (Experimental): A heart ultrasound using a handheld ultrasound device will be used during a pacemaker implant procedure
  Interventions: Device: Heart Ultrasound

INTERVENTIONS:
Device: Heart Ultrasound — A wand is placed on the chest to use soundwaves to make a picture of the heart and shows how the muscle and valves work. This helps with device placement.
  Arms: EC-LBBAP Participant; ECLBBAP handheld participant

SUMMARY:
The goal of this observational study is to learn more about whether or not the use of heart ultrasound during pacemaker implantation is helpful. The main questions this aims to answer are:

1. Does this help the doctors with figuring out the wire location during implantation?
2. Does this reduce the wire placement procedure time?
3. Does this reduce the x-ray imaging time during the procedure?

Participants will be asked to:

1. Have a physical exam and Echocardiogram (ECG) at initial visit, 2 weeks post implant, and 3 months post implant.
2. Have a urine pregnancy test (if applicable)
3. Have a heart ultrasound during implant procedure
4. Answer questions related to heart failure symptoms to see what stage of heart failure is present
5. Have device interrogation (a wand placed over the chest to see that the device is working properly) at a visit 2 weeks post implant and at 3 months post implant.

DETAILED DESCRIPTION:
The EC-LBBAP study is a prospective, single-enter, observational research study. The study team will identify all patients who satisfy the inclusion and exclusion criteria. The study team will evaluate the feasibility and success rates of echocardiogram guided LBBAP lead implantation.

Eligible patients will undergo LBBAP using Medtronic 3830 lead and C315His sheath. LBBAP will be confirmed at implant using left bundle potentials recorded from the lead, ECG morphology during unipolar and bipolar pacing, peak Left Ventricular Pacing (LV) activation time and lead depth in the 2D transthoracic echo at implant.

During implant procedure, transthoracic echo windows will be identified and documented: Parasternal short and long axis, apical 2 and 4 chamber views and subcostal views to visualize the proximal interventricular septum. Following venous access using cephalic vein cut-down or ultrasound guided axillary vein access, the lead implantation in the left bundle branch region will be guided by echocardiography.

Retrospectively, the study team will identify 20 consecutive previous patients who satisfy inclusion and exclusion criteria (control patients). Twenty patients will undergo intraprocedural transthoracic echocardiogram via standard practices. An additional 10 patients will undergo intraprocedural transthoracic echocardiogram using a hand-held ultrasound device. The study team will compare the difference in procedural success between case and control patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with indication for permanent pacemaker or Implantable Cardioverter Defibrillator (ICD) utilizing conduction system pacing lead for bradycardia or cardiac resynchronization therapy
* patient is willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Inability to provide informed consent
* pregnant
* enrolled in a concurrent study that may confound the results of this study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pugazhendhi Vijayaraman, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared in an identifiable way.

REFERENCES:
- [Derived] Vijayaraman P, Hughes G, Manganiello M, Leri G, Laver A, Sacco K, Mroczka K, Schmidt E, Mascarenhas VH. Intraprocedural transthoracic EChocardiography to facilitate Left Bundle Branch Pacing: EC-LBBP. Heart Rhythm. 2025 Sep;22(9):e746-e753. doi: 10.1016/j.hrthm.2024.12.039. Epub 2024 Dec 31. PMID 39746387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants will be identified by clinician referrals at Geisinger Wyoming Valley Heart Hosptial. Research staff will contact potential subjects and invite them to participate.
Pre-assignment Details: 21 EC-LBBAP participants were consented and enrolled in the study. One participant did not complete the study and was exited, as echo was unable to be complete at implant.
  12 EC-LBBAP handheld participants were consented and enrolled in the study. Two participants did not complete the study and were exited, as echo was unable to be complete at implant.
  30 Participants in the "Control" Arm/Group are not considered enrolled and therefore, not included in the Number Enrolled.
Period: Overall Study
Arm/Group | EC-LBBAP Participant | Control Participant | ECLBBAP Handheld Participant
Started | 21 | 30 | 12
Completed | 20 | 30 | 10
Not Completed | 1 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EC-LBBAP Participant | Control Participant | ECLBBAP Handheld Participant | Total
Number analyzed (Participants) | 20 | 30 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Age
  years | 71.35 (10.236) | 77.06 (9.18) | 72.8 (12.5) | 74.45 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 4 | 25
  Male | 10 | 19 | 6 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 28 | 10 | 58
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (5.63) | 28.74 (5.27) | 26.9 (6.48) | 28.8 (5.58)
Hypertension [Count of Participants; unit: Participants] | 17 | 28 | 10 | 55
Diabetes [Count of Participants; unit: Participants] | 5 | 10 | 5 | 20
Coronary artery disease [Count of Participants; unit: Participants] | 9 | 12 | 3 | 24
Atrial Fibrillation [Count of Participants; unit: Participants] | 15 | 21 | 5 | 41
Cardiomyopathy [Count of Participants; unit: Participants] | 7 | 21 | 5 | 33

OUTCOME MEASURES:

1. Primary Outcome: A Positive Success Rate of LBBAP Utilization With Intraprocedural Transthoracic Echocardiogram
Description: Positive success rate of LBBAP is measured by Left bundle branch capture for participants, measured during implant
Time Frame: Perioperative, through study completion, an average of 3 months
Measure: Count of Participants; unit: Participants
Groups:
- EC-LBBAP Participant: Patients undergoing pacemaker insertion using ultrasound guided left bundle branch pacing
- EC-LBBAP Handheld Participant: Patients undergoing pacemaker insertion using handheld ultrasound guided left bundle branch pacing
Arm/Group | EC-LBBAP Participant | EC-LBBAP Handheld Participant
Number analyzed (Participants) | 20 | 10
Participants | 19 | 10

2. Primary Outcome: Difference of Fluoroscopy/Procedure Duration Between Groups
Description: Difference in fluoroscopy and procedure duration using echo guided LBBAP lead implantation compared to control data for standard LBBAP lead implantation
Time Frame: Perioperative
Measure: Median (Standard Deviation); unit: min
Groups:
- Standard LBBP: Patients undergoing pacemaker insertion using standard practice for left bundle branch pacing
Arm/Group | EC-LBBAP Participant | EC-LBBAP Handheld Participant | Standard LBBP
Number analyzed (Participants) | 20 | 10 | 30
min
  Procedure duration | 101 (27) | 89 (29) | 95 (39)
  Fluoroscopy duration | 8.9 (7.9) | 10.1 (6.5) | 13.5 (8.5)

3. Primary Outcome: Number of Participants Determined to be Eligible for the Work-flow and Echocardiographic Procedures
Description: This measure is to determine if the workflow is feasible in regular practice (echo tech availability, lab availability, duration of comparative procedures) between intervention group and controls, and to determine if the identifying echocardiographic windows is able to be performed pre operatively on all intervention patients
  This measure is to determine the number of participants that the workflow is feasible for and could be performed on in regular practice (echo tech availability, lab availability, duration of comparative procedures)
Time Frame: Through study completion, an average of 3 months
Population: Workflow defined and echo images obtained to facilitate LBBAP in participants in the ECLBBAP arm
Measure: Number; unit: participants
Arm/Group | EC-LBBAP Participant | EC-LBBAP Handheld Participant
Number analyzed (Participants) | 20 | 10
participants | 20 | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected during study participation up to final study visit at 3 months post implant.
Description: Patients will be asked about adverse events related to the use of the echocardiography. Only echocardiogram related adverse event will be collected and reported and then assessed if it is procedure related, as well as all-cause mortality and serious adverse events.
Arm/Group | EC-LBBAP Participant | Control Participant | ECLBBAP Handheld Participant
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT05646251/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT05646251/ICF_001.pdf